CLINICAL TRIAL: NCT01807117
Title: Evaluation of PET-MRI in Initial Staging of High Grade Rectal Cancer Patients and in the Follow up of Colorectal Cancer Patients.
Brief Title: PET-MRI in Diagnosing Patients With Colon or Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CASE8212; NCI-2013-00511 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-03-06; First posted 2013-03-08 (Estimated); Results first posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-04

CONDITIONS: Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage IIA Colon Cancer; Stage IIA Rectal Cancer; Stage IIB Colon Cancer; Stage IIB Rectal Cancer; Stage IIC Colon Cancer; Stage IIC Rectal Cancer; Stage IIIA Colon Cancer; Stage IIIA Rectal Cancer; Stage IIIB Colon Cancer; Stage IIIB Rectal Cancer; Stage IIIC Colon Cancer; Stage IIIC Rectal Cancer; Stage IVA Colon Cancer; Stage IVA Rectal Cancer; Stage IVB Colon Cancer; Stage IVB Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (PET-CT and PET-MRI) (Experimental): Patients undergo fludeoxyglucose F 18 PET-CT and PET-MRI.
  Interventions: Procedure: positron emission tomography; Procedure: computed tomography; Procedure: magnetic resonance imaging; Radiation: fludeoxyglucose F 18

INTERVENTIONS:
Procedure: positron emission tomography — Undergo fludeoxyglucose F 18 PET-CT and PET-MRI
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Procedure: computed tomography — Undergo fludeoxyglucose F 18 PET-CT and PET-MRI
  Other Names: tomography, computed
Procedure: magnetic resonance imaging — Undergo fludeoxyglucose F 18 PET-CT and PET-MRI
  Other Names: MRI; NMR imaging; NMRI; nuclear magnetic resonance imaging
Radiation: fludeoxyglucose F 18 — Undergo fludeoxyglucose F 18 PET-CT and PET-MRI
  Other Names: 18FDG; FDG

SUMMARY:
This pilot clinical trial studies positron emission tomography (PET)-magnetic resonance imaging (MRI) and PET-computed tomography (CT) as diagnostic imaging in patients with colon and/or rectal cancer. New diagnostic imaging procedures, such as PET-MRI, may help find and diagnose rectal cancer or recurrence of colorectal cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test the diagnostic performance of PET- MRI in the staging of preoperative high-grade rectal cancer patients, defined by T3 stage or higher or N1 stage or higher or presence of metastasis, that are referred to PET-CT and MRI.

II. To test the diagnostic performance of PET-MRI the follow up of colorectal cancer patients that are referred to PET-CT with or without a diagnostic MRI request by their physicians.

SECONDARY OBJECTIVES:

I. To test different attenuation correction MR sequences and novel diagnostic MR sequences.

OUTLINE:

Patients undergo fludeoxyglucose F 18 PET-CT and PET-MRI.

ELIGIBILITY:
Inclusion Criteria:

* Either having a T3 (the cancer has grown through the muscularis propria and into the outermost layers of the colon or rectum but not through them) or higher, node positivity or metastatic lesion in the context of rectal cancer or being studied for colorectal cancer follow up, independent of the renal function
* PET-CT should be requested by a referring physician; in the case of having an MR requested as well, it will be reported from the MRI images generated in the PET-MRI
* Stable physical medical conditions to undergo a MRI
* Informed consent must be given and signed prior to study enrollment

Exclusion Criteria:

* Refuse to give and/or sign the informed consent
* Subjects who do not meet the above mentioned inclusion criteria
* Subjects who have a pacemaker
* Subjects who have a metallic prostheses either in the pelvis or in the abdomen that will interfere with the MR imaging of that anatomical area
* Subjects who suffer from claustrophobia
* Pregnant women
* Cognitive impairment that affects the subject's ability to give consent

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2014-03-05 (Actual); Study Completion 2014-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raj Paspulati, MD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diagnostic (PET-CT and PET-MRI)
Started | 15
Completed | 12
Not Completed | 3
Not completed — Physician Decision | 2
Not completed — Disease diagnosis not a study disease | 1

BASELINE CHARACTERISTICS:
Population: Participants who were put on study
Arm/Group | Diagnostic (PET-CT and PET-MRI)
Number analyzed (Participants) | 15
Age, Customized [Count of Participants; unit: Participants]
  years: 20-29 | 0
  years: 30-39 | 0
  years: 40-49 | 4
  years: 50-59 | 3
  years: 60-69 | 4
  years: 70-79 | 4
  years: 80-89 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 0
  More than one race | 8
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Maximum Standardized Uptake Value (SUVmax) in Physiologic Regions and Fluorodeoxyglucose (FDG) Avid Lesions in Participants Where PET-CT Was Performed Prior to the PET-MRI
Description: SUV max in physiologic regions (blood pool, liver) and FDG avid lesions, in which the PET-CT was performed prior to the PET-MRI. SUVmax is defined as [tissue concentration (MBq/g) x body weight (g)]/[injected dose (MBq/g)]
Time Frame: Up to 6 months (each scan taking an average of 45 minutes)
Population: Participants who received PET-CT as initial imaging followed by PET-MRI. Evaluable lesions for this group.
Measure: Median (Full Range); unit: SUV max
Units Other Than Participants: Lesions
Groups:
- Blood Pool: Physiologic region - Diagnostic (PET-CT and PET-MRI) arm
  Patients undergo fludeoxyglucose F 18 PET-CT and PET-MRI.
  positron emission tomography: Undergo fludeoxyglucose F 18 PET-CT and PET-MRI
  computed tomography: Undergo fludeoxyglucose F 18 PET-CT and PET-MRI
  magnetic resonance imaging: Undergo fludeoxyglucose F 18 PET-CT and PET-MRI
  fludeoxyglucose F 18: Undergo fludeoxyglucose F 18 PET-CT and PET-MRI
- Liver: Physiologic region - Diagnostic (PET-CT and PET-MRI) arm Physiologic region - Diagnostic (PET-CT and PET-MRI) arm
  Patients undergo fludeoxyglucose F 18 PET-CT and PET-MRI.
  positron emission tomography: Undergo fludeoxyglucose F 18 PET-CT and PET-MRI
  computed tomography: Undergo fludeoxyglucose F 18 PET-CT and PET-MRI
  magnetic resonance imaging: Undergo fludeoxyglucose F 18 PET-CT and PET-MRI
  fludeoxyglucose F 18: Undergo fludeoxyglucose F 18 PET-CT and PET-MRI
Arm/Group | Blood Pool | Liver
Number analyzed (Participants) | 9 | 9
Number analyzed (Lesions) | 23 | 23
SUV max
  PET-CT | 1.9 [1.2 to 2.5] | 2.3 [1.7 to 3.4]
  PET-MRI | 1.3 [0.8 to 1.6] | 2.1 [1.6 to 3.4]

2. Primary Outcome: Maximum Standardized Uptake Value (SUVmax) in Physiologic Regions and FDG Avid Lesions in Participants Where PET-MRI Was Performed Prior to the PET-CT
Description: SUV max in physiologic regions (blood pool, liver) and FDG avid lesions, in which the PET-MRI was performed prior to the PET-CT. SUVmax is defined as [tissue concentration (MBq/g) x body weight (g)]/[injected dose (MBq/g)]
Time Frame: Up to 6 months (each scan taking an average of 45 minutes)
Population: Participants who received PET-MRI was performed prior to the PET-CT. Evaluable lesions for this group.
Units Other Than Participants: Lesions
Arm/Group | Blood Pool | Liver
Number analyzed (Participants) | 0 | 0
Number analyzed (Lesions) | 0 | 0

3. Primary Outcome: SUVmax in Which the PET-CT Was Performed Prior to the PET-MRI.
Description: SUVmax in FDG avid lesions in which the PET/CT was performed prior to the PET-MRI.
  SUVmax is defined as [tissue concentration (MBq/g) x body weight (g)]/[injected dose (MBq/g)]
Time Frame: Up to 6 months (each scan taking an average of 45 minutes)
Population: Participants who received PET-CT as initial imaging followed by PET-MRI. Evaluable lesions for this group.
Measure: Median (Full Range); unit: SUV max
Units Other Than Participants: Lesions
Arm/Group | Diagnostic (PET-CT and PET-MRI)
Number analyzed (Participants) | 9
Number analyzed (Lesions) | 16
SUV max
  PET-CT | 3.0 [0.5 to 25.5]
  PET-MRI | 3.9 [1.6 to 21.6]

4. Primary Outcome: SUVmax in Which the PET-MRI Was Performed Prior to the PET-CT
Description: SUVmax in FDG avid lesions in which the PET-MRI was performed prior to the PET-CT SUVmax is defined as [tissue concentration (MBq/g) x body weight (g)]/[injected dose (MBq/g)]
Time Frame: Up to 6 months (each scan taking an average of 45 minutes)
Population: Participants who received PET-MRI as initial imaging followed by PET-CT. Evaluable lesions for this group.
Measure: Median (Full Range); unit: SUV max
Units Other Than Participants: Lesions
Arm/Group | Diagnostic (PET-CT and PET-MRI)
Number analyzed (Participants) | 3
Number analyzed (Lesions) | 7
SUV max
  PET-CT | 5.9 [3.4 to 8.0]
  PET-MRI | 4.3 [2.3 to 6.3]

5. Primary Outcome: SUVmax Ratio in Which the PET-CT Was Performed Prior to the PET-MRI
Description: SUVmax ratio in FDG avid lesions in which the PET-CT was performed prior to the PET-MRI
  SUVmax is defined as [tissue concentration (MBq/g) x body weight (g)]/[injected dose (MBq/g)]
Time Frame: Up to 6 months (each scan taking an average of 45 minutes)
Population: Participants who received PET-CT as initial imaging followed by PET-MRI. Evaluable lesions for this group.
Measure: Median (Full Range); unit: SUV max ratio
Units Other Than Participants: Lesions
Arm/Group | Diagnostic (PET-CT and PET-MRI)
Number analyzed (Participants) | 9
Number analyzed (Lesions) | 16
SUV max ratio
  PET-CT | 2.0 [0.2 to 11.1]
  PET-MRI | 2.5 [0.8 to 10.8]

6. Primary Outcome: SUVmax Ratio in Which the PET-MRI Was Performed Prior to the PET-CT
Description: SUVmax ratio in FDG avid lesions in which the PET-MRI was performed prior to the PET-CT SUVmax is defined as [tissue concentration (MBq/g) x body weight (g)]/[injected dose (MBq/g)]
Time Frame: Up to 6 months (each scan taking an average of 45 minutes)
Population: Participants who received PET-MRI as initial imaging followed by PET-CT. Evaluable lesions for this group.
Measure: Median (Full Range); unit: SUV max
Units Other Than Participants: Lesions
Arm/Group | Diagnostic (PET-CT and PET-MRI)
Number analyzed (Participants) | 3
Number analyzed (Lesions) | 7
SUV max
  PET-CT | 2.7 [1.5 to 7.2]
  PET-MRI | 2.0 [1.2 to 7.0]

7. Primary Outcome: True Positive Rate
Description: True positive rate for both modalities - TP/TP+FN
  TP = true positives FN = False negatives
Time Frame: Up to 6 months (each scan taking an average of 45 minutes)
Population: Evaluable lesions for this group.
Measure: Number; unit: percentage of true positive results
Units Other Than Participants: Lesions
Arm/Group | Diagnostic (PET-CT and PET-MRI)
Number analyzed (Participants) | 12
Number analyzed (Lesions) | 23
percentage of true positive results
  PET-CT | 71
  PET-MRI | 71

8. Primary Outcome: True Negative Rate
Description: True negative rate for both modalities - TN/TN+FP
  TN = true negatives FP = False positives
Time Frame: Up to 6 months (each scan taking an average of 45 minutes)
Measure: Number; unit: percent
Units Other Than Participants: Lesions
Arm/Group | Diagnostic (PET-CT and PET-MRI)
Number analyzed (Participants) | 12
Number analyzed (Lesions) | 23
percent
  PET-CT | 100
  PET-MRI | 100

9. Primary Outcome: False Negative Rate
Description: False negative rate for both modalities - FN/FN+TP
  FN = False negatives TP = true positives
Time Frame: Up to 6 months (each scan taking an average of 45 minutes)
Population: Evaluable lesions for this group.
Measure: Number; unit: percent
Units Other Than Participants: Lesions
Arm/Group | Diagnostic (PET-CT and PET-MRI)
Number analyzed (Participants) | 12
Number analyzed (Lesions) | 23
percent
  PET-CT | 29
  PET-MRI | 14

10. Primary Outcome: Proportion of Lesions Identified by PET-CT That Were Correctly Detected by PET-MRI
Description: On a per-lesion basis, proportion of lesions identified by PET-CT that were correctly detected by PET-MRI
Time Frame: Up to 6 months (each scan taking an average of 45 minutes)
Measure: Number; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Diagnostic (PET-CT and PET-MRI)
Number analyzed (Participants) | 12
Number analyzed (Lesions) | 29
Lesions | 26

11. Primary Outcome: Positive Predictive Values for PET-CT and PET-MRI
Description: Percent of true positive rate of diagnostic accuracy.
Time Frame: Up to 6 months (each scan taking an average of 45 minutes)
Population: Evaluable lesions for this group.
Measure: Number; unit: Percent of true positives
Units Other Than Participants: Lesions
Arm/Group | Diagnostic (PET-CT and PET-MRI)
Number analyzed (Participants) | 12
Number analyzed (Lesions) | 23
Percent of true positives
  PET-CT | 100
  PET-MRI | 100

12. Primary Outcome: Negative Predictive Values for PET-CT and PET-MRI
Description: Percent of true negative rate of diagnostic accuracy
Time Frame: Up to 6 months (each scan taking an average of 45 minutes)
Population: Evaluable lesions for this group.
Measure: Number; unit: Percent of true negatives
Units Other Than Participants: Lesions
Arm/Group | Diagnostic (PET-CT and PET-MRI)
Number analyzed (Participants) | 12
Number analyzed (Lesions) | 23
Percent of true negatives
  PET-CT | 71.43
  PET-MRI | 83.33

ADVERSE EVENTS:
Time Frame: Adverse events: At time of intervention, an average of 1 hour Survival: Up to 5 years
Arm/Group | Diagnostic (PET-CT and PET-MRI)
All-Cause Mortality (participants affected / at risk) | 6/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-10-18): https://cdn.clinicaltrials.gov/large-docs/17/NCT01807117/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-16): https://cdn.clinicaltrials.gov/large-docs/17/NCT01807117/ICF_001.pdf